CLINICAL TRIAL: NCT03189238
Title: A Double Blind Placebo Controlled Trial of Autologous Platelet Rich Plasma (PRP) Peri-urethral and Clitoral Injections for the Treatment of Female Orgasmic Disorder
Brief Title: Platelet Rich Plasma (PRP) Peri-urethral and Clitoral Injections for the Treatment of Female Orgasmic Disorder
Acronym: PRP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Vulvovaginal Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00021800
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Female Orgasmic Disorder

STUDY DESIGN:
Intervention Model Description: This will be a single center study with 40 female patients; twenty placebo and twenty active treatment patients.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: Peri-urethral and clitoral injections
- PRP (Active Comparator)
  Interventions: Biological: Peri-urethral and clitoral injections

INTERVENTIONS:
Biological: Peri-urethral and clitoral injections — Peri-urethral and clitoral injections

SUMMARY:
Female Orgasmic Disorder (FOD) is defined as a female sexual disorder with the presence of the following "on all or almost all (75%-100%) occasions of sexual activity":

1. Marked delay in, marked infrequency of, or absence of orgasm
2. Marked reduced intensity of orgasmic sensations.
3. The absence of orgasm must cause personal distress (bother) in order for these symptoms to be considered a disorder. (for example, women who are not very bothered by their lack of orgasm do not have FOD).

Symptoms must have been present for at least 6 months and are not better explained by a mental disorder or because of a relationship problems or other significant stress in the participant's life and not due to effects of substance abuse or new medications or other medical conditions.

Approximately one in twenty women have FOD and it is the second most frequently reported sexual problem in American women. FOD can either be lifelong (primary) or acquired (secondary).

There are no currently FDA approved treatments or devices for FOD. Therefore, common off-label treatments include psychotherapy/sex therapy, hormone therapy, and medications that increase blood flow to the genitals.

Platelet-rich plasma (PRP) is a platelet concentrate that may help to speed up tissue healing, without serious side effects, in some medical conditions. It has been tried as treatment for diabetic foot ulcers, muscle injury, tendon injury, and in a variety of cosmetic procedures. The only condition for which there are high-quality data and clear demonstration of effectiveness is arthritis of the knee. It is also apparent from the majority of published studies that PRP therapy has minimal risk of scar tissue formation or significant bad side effects.

It has been suggested by many scientists that in some women FOD may be caused by decreased clitoral and genital blood flow secondary to blockage in the small blood vessels going to the clitoris (similar to that seen in erectile dysfunction (ED) in men) and/or diminished nerve conduction (also as seen in ED). PRP activates cells to develop into new tissue-nerves, collagen, and blood vessels. As such, PRP may potentially reverse the changes responsible for FOD. In addition, it has been shown that improved sexual function in women is highly linked with increased blood flow through the clitoris. One component of PRP is known to cause growth of new blood vessels. Therefore, the investigators anticipate PRP injections may potentially improve blood flow through both the clitoris and the tissue around the urethra, thereby improving sexual function and decreasing FOD.

In addition, it has been shown that women who easily achieve orgasm are more likely than women with FOD to have a larger clitoris and a clitoris positioned closer to the vaginal wall. Since PRP has been shown to increase connective tissue, injection of PRP into the clitoris may potentially enlarge the clitoris and may bring the clitoris closer to the vaginal wall, thereby improving orgasm.

There are some reports that physicians using the PRP as an injection near the urethra and clitoris have seen some patients with improvement in FOD after the injections. This is the first study that uses an objective comparative study to find out if this treatment works or not.

ELIGIBILITY:
Inclusion Criteria:

< Female, 25-50 years old. < Premenopausal < Signed written informed consent. < Willingness and ability to comply with the study requirements. < Subject must meet all of the criteria of FOD as listed in the DSM 5 < Subjects must score between 0-4 on the Orgasm Domain of the FSFI < Previously had satisfying orgasms < Score 11 or greater on the Female Sexual Distress Scale - revised (FSDS-R) < Are in a continuous, stable sexual relationship with the same partner for at least the 12 months immediately before study enrollment

Exclusion Criteria:

< Who are menopausal < Who have primary FOD < Who have pain during sex < Who are immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have an uncontrolled malignant disease.

< Who are not in a stable sexual relationship of at least 12 month duration < Who suffer from systemic or generalized infections (bacterial, viral or fungal).

< Taking psychotropic medications including SSRIs, SNRIs, TCA, bupropion, mood stabilizers, & treatments for ADD or ADHD including Adderall and similar compounds.

< Taking sildenafil, vardenafil, tadalafil < Taking topical or systemic estrogen or testosterone < Taking oral contraceptive pills < Who have been diagnosed with lichen sclerosus, lichen planus, psoriasis, candidiasis, intraepithelial neoplasia, or carcinoma of the vulva.

< Who had received an investigational drug within four weeks prior to the study or who intend to use other investigational drugs during the course of this study.

< Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.

< Who have a history of substance abuse or any factor, which limits the subject's ability to cooperate with the study procedures.

Who are uncooperative, known to miss appointments (according to subjects' records) and are unlikely to follow medical instructions or are not willing to attend regularly scheduled visits.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-28 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
ANCOVA | 2 months
  The ANCOVA will give the investigators adequate power for the proposed sample size (20+20). From the reports of clinicians performing the treatment, the investigators are estimating that the effects to be significant for about 80% of clients. The placebo effect for sexual dysfunction is usually around 40% (see Bradford review, 2013) so that the estimated difference is 40 points which corresponds to a RR (risk ration) = 2, a large effect. A repeated measure ANCOVA with 20 participants per group (2 groups) would have 80% chance of finding a significant difference between groups if the effect size was at least d = .88. An 80% chance is a standard experimental choice that is in line with clinical and medical trials. A Cohen's d above .8 is considered large effect for a treatment study and a d between .5 and .8 is considered medium, thus a sample of 20 + 20 participants is estimated to be adequate to find a large effect as the one expected for this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Goldstein, MD, Principal Investigator — Director
Locations (1):
- The Center for Vulvovaginal Disorders, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Informed Consent Form — http://cvvd.org/research — Link for the informed consent is in the section titled "PLATELET RICH PLASMA (PRP) INJECTIONS FOR THE TREATMENT OF FEMALE ORGASMIC DISORDER."